CLINICAL TRIAL: NCT00580437
Title: The Analysis of Data Collected During Angiography and Dobutamine Stress Contrast Echocardiograms in the Pre-Evaluation of Kidney and Pancreas Transplant Patients
Brief Title: Pre-operative Evaluation of Kidney & Pancreas Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0142-03-EP
Record Dates: First submitted 2007-12-17; First posted 2007-12-24 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplantation; Pancreas Transplantation
MeSH Terms: interventions — perflutren; FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): stress echocardiograms involving the use of intravenous Optison or Definity contrast agents to improve endocardial definition
  Interventions: Procedure: Dobutamine Stress Echocardiogram

INTERVENTIONS:
Procedure: Dobutamine Stress Echocardiogram — stress echocardiograms involving the use of intravenous Optison or Definity contrast agents to improve endocardial definition
  Other Names: Definity; Optison

SUMMARY:
Examine the clinical utility of the dobutamine stress contrast echoes and angiograms obtained routinely in the evaluation of patients prior to kidney or pancreas transplantation.

DETAILED DESCRIPTION:
Although there is an increasing quantity of data demonstrating the value of stress echo in risk stratifying patients for cardiac risk prior to major non-cardiac surgery, the current clinical practice utilized for assessing patients being evaluated for kidney or pancreas transplantation is both a stress echocardiogram and a coronary angiogram. This gap in opinion appears to be a concern on the part of both nephrologists, endocrinologists, and surgeons that the stress echocardiogram may miss significant angiographic disease that could result in major post-operative complications in this high-risk subgroup of patients (unstable angina, non-fatal infarction, or death).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are being evaluated for a kidney and or pancreas transplant and scheduled for a dobutamine stress echocardiogram and a coronary angiogram will be eligible to participate

Exclusion Criteria:

* Patients with unstable angina at the time of their evaluation, or who have a severe underlying cardiomyopathy or valve disease will be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-05-02 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2012-04-01 (Actual)

PRIMARY OUTCOMES:
Stress echocardiogram diagnostic sensitivity | prior to transplantation
  Prior to the pancreas or kidney transplant, wall motion by stress echocardiograms indicates the cardiac risk. Intravenous administered Optison or Definity contrast agents during the stress echo improve endocardial definition, enabling better assessment of myocardial perfusion and significant angiographic disease. This is particularly crucial in the high-risk subgroup of patients (unstable angina, non-fatal infarction, or death) to identify potential major post-operative complications.
Event-free survival | 3 years
  Patients were followed up for the primary outcome variable, event-free survival (EFS), defined as the time from transplant to the incidence of myocardial infarction, heart failure hospitalization, or all-cause mortality. Analyze EFS in pancreas or kidney transplant patients.

SECONDARY OUTCOMES:
Abnormal stress myocardial perfusion rate | 3 years
  Analyze myocardial perfusion simultaneously during the replenishment phase of contrast following high mechanical index impulses using a 17-segment model. Any abnormal perfusion response had to be confirmed by a second independent expert reviewer, blinded to angiographic or clinical outcome data. Fixed or inducible segments were considered abnormal. Calculate the abnormal stress myocardial perfusion rate in the transplant patients and analyze the association with the risk of an event after transplantation.
Abnormal stress wall motion rate | 3 years
  Analyze wall motion simultaneously during the replenishment phase of contrast following high mechanical index impulses using a 17-segment model. Any abnormal wall motion response had to be confirmed by a second independent expert reviewer, blinded to angiographic or clinical outcome data. Fixed or inducible segments were considered abnormal. Calculate the abnormal stress wall motion rate in the transplant patients and analyze the association with the risk of an event after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Porter, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States